## CONSENT BY PATIENT FOR CLINICAL RESEARCH

| I, | |
|---|---|
| Identity Card No | |
| (Name of Patient) | |
| of | duaga) |
| | dress) |
| below: | linical study/questionnaire study/drug trial) specified |
| <u>Title of Study:</u> <i>Lignosus rhinocerus</i> TM02® as an in uncontrolled asthma: A prospective, open-label, Pha | |
| the nature and purpose of which has been explained to me by Dr | |
| (Name & Designation of Doctor) and interpreted by | |
| (Name & Designation of Interpreter) | |
| to the best clanguage/dialect. | of his/her ability in |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. | |
| | l research at any time without assigning any reason<br>nied the benefits of usual treatment by the attending |
| Date: Signature or | Thumbprint |
| (Patient) | |
| IN THE PRESENCE OF | |
| Name) | |
| Identity Card No | Signature |
| | (Witness for Signature of Patient) |
| Designation) | (withess for signature of Lutterit) |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. | |
| Date | Signature(Attending Doctor) |
| CONSENT BY PATIENT R.N. FOR Name | |
| CLINICAL RESEARCH Sex | |
| Age | |
| I Unit | |

## CONSENT BY RESPONSIBLE RELATIVE FOR CLINICAL RESEARCH

| I, | | |
|---|---|---|
| Identity Card No | | |
| of(Name) | | |
| of | dress) | |
| (Au | uress) | |
| hereby agree that my relative | | |
| I.C. No(Name) | | |
| participate in the clinical research (clinical stud | dy/question | naire study/drug trial) specified below:- |
| <u>Title of Study:</u> <i>Lignosus rhinocerus</i> TM02® auncontrolled asthma: A prospective, open-lal | | |
| the nature and purpose of which has been exp | lained to m | e by Dr. |
| (Name & Designation of Doctor) | | |
| and interpreted by(Name & Designation | of Interpret | <br>2r) |
| to the best of his | s/her ability | inlanguage/dialect. |
| and complications (as per patient informa | tion sheet) | h in terms of procedure, possible adverse effects . I understand the possible advantages and rily give my consent for my relative to participate |
| reason whatsoever and in such situation, my r | elative shall<br>gains his/he | inical research at any time without assigning any not be denied the benefits of usual treatment by r ability to consent, he/she will have the right to |
| Relationship Date: to Patient | | Signature or Thumbprint |
| IN THE PRESENCE OF | | |
| Name) | 1 | |
| Identity Card No | )<br>) | Signature( <i>Witness</i> ) |
| Designation) | , | (WithEss) |
| I confirm that I have explained to the patient's clinical research. | relative the | nature and purpose of the above-mentioned |
| Date | | Signature(Attending Doctor) |
| R.N. | | |
| CONSENT BY<br>RESPONSIBLE RELATIVE FOR<br>CLINICAL RESEARCH | Name<br>Sex<br>Age | Unit |

BK-MIS-1117-E01 Version 1.0 dated 23 OCT 2020